CLINICAL TRIAL: NCT06793306
Title: A Study Comparing the Differences Between Young and Non-young Breast Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, PENG YUAN, Head of department, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC5093
Record Dates: First submitted 2025-01-18; First posted 2025-01-27 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Aging; Combined Modality Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Breast cancer
  Interventions: Other: Age; Other: combination therapy

INTERVENTIONS:
Other: Age — Breast cancer patients were divided into young breast cancer and non-young breast cancer by age 35
Other: combination therapy — To observe and compare the difference in diagnosis, combined treatment and prognosis between young and non-young breast cancer

SUMMARY:
To collect data on diagnosis, treatment, survival prognosis, and intrinsic molecular detection of breast cancer in China from January 2000 to December 2024.Compare the difference between young and non-young breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* During the period from January 2000 to December 2024, the first breast cancer diagnosed and treated in several hospitals in China was in the age range of 18-75 years.

Exclusion Criteria:

* Breast cancer patients under 18 years of age or over 75 years of age; Combined with other malignant tumors; Patients with chronic infectious diseases or chronic infectious diseases; Patients with severe comorbidities, with serious dysfunction of vital organs (heart, liver, kidney); Known history of human immunodeficiency virus; The investigator concluded that patients should not be included in other conditions of this trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During the period from January 2000 to December 2024, the first breast cancer diagnosed and treated in several hospitals in China was in the age range of 18-75 years. Young patients with breast cancer were defined as ≤35 years old, and non-young patients were defined as patients over 35 years old.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 10-year

SECONDARY OUTCOMES:
invasive disease-free survival rate | 10-year

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No